CLINICAL TRIAL: NCT01050010
Title: The Relation Between Dedicated Extremity MRI Synovitis and Structural Deterioration Radiographic in Patients With Rheumatoid Arthritis in Clinical Remission.Preliminary Study
Brief Title: The Relation Between Dedicated Extremity MRI Synovitis and Structural Deterioration Radiographic in Patients With Rheumatoid Arthritis in Clinical Remission. Preliminary Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 09-CIR-01
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; clinical remission; synovitis; dedicated extremity MRI
MeSH Terms: conditions — Arthritis, Rheumatoid; Synovitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dedicated extremity MRI (Other): Structural deterioration radiographic assessed by dedicated extremity MRI
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — dedicated extremity MRI

SUMMARY:
The major aim of treatment for rheumatoid arthritis is remission. Nevertheless, structural radiographic progression is observed in 15 to 20% of patient getting remission. Numerous definitions of the remission proposed by literature remain imperfect.

Recently ultrasonography and MRI seem to be helpful in diagnosis and follow-up of rheumatoid arthritis.

Studies in patients with clinical remission are reporting 75 to 90% of persistent MRI and ultrasonography synovitis, 45% of cases with synovial activity.

To our knowledge, in such case few studies showed correlation between persistent imaging synovitis and structural radiographic progression.

On the other hand, no studies with extremity dedicated RMI in patients with remission are reported.

In this preliminary study, the investigators propose to evaluate in patients with rheumatoid arthritis remission and persistent dedicated MRI synovitis the structural radiographic progression at one year.

ELIGIBILITY:
Inclusion Criteria:

* Earlier rheumatoid arthritis (<1 year)
* Clinical remission (DAS 28 <2,6 ou SDAI <5) since 6 months before the inclusion
* Unchanged DMARds and /or biologic therapy since 6 months before the inclusion
* Unchanged corticosteroid (5 mg/day) since 3 months before the inclusion in patients treated with this therapy
* No contre-indication to the MRI

Exclusion Criteria:

* Contra-indication to MRI
* Pregnant or breast-feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Dedicated extremity MRI (hand and wrist)/ X-Ray (hand, wrist and foot) | at Month 0 (first visit) and Month 12 (last visit)

SECONDARY OUTCOMES:
Ultrasonography (hand, wrist and foot) | at Month 0 (first vist) and Month 12 (last visit)

CONTACTS AND LOCATIONS:
Overall Officials: Christine ALBERT-SABONNADIERE, PhD, Principal Investigator — Nice University Hospital
Locations (2):
- France (2):
  - CHU de NICE, Nice
  - Rheumatology Department, Nice University Hospital, Nice